CLINICAL TRIAL: NCT02340663
Title: Preliminary Phase IV Trial Comparing the SOVA Night Guard With the Clinical Standard Acrylic Orthotic
Brief Title: Nocturnal Mouth Guards, SOVA vs. Standard Acrylic Orthotic; Phase IV
Acronym: SISU-SOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Delta Dental Fund of Michigan (Other)
Responsible Party: Principal Investigator, Geoffrey E. Gerstner, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00085489
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Sleep Bruxism; Tooth Wear
Keywords: dental orthotic; bite splint; oral parafunction; clenching; grinding
MeSH Terms: conditions — Sleep Bruxism; Tooth Wear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOVA bite splint (Experimental): SOVA Bite splint: Over-the-counter, heat-and-mold bite splint. Investigators evaluate subject self-fabrication, and evaluate fit. Subjects wear splint nightly for one week. Polysomnographic data obtained from one night during the week. Subjects continue to wear splint for 3 months, dairy kept of nightly wear. Polysomnographic data obtained from one night at the end of three months.
  Interventions: Device: SOVA Bite Splint
- Michigan Bite Splint (Active Comparator): Michigan bite splint: Gold standard, custom acrylic bite splint made for subjects. Investigators evaluate fit. Subjects wear splint nightly for one week. Polysomnographic data obtained from one night during the week. Subjects continue to wear splint for 3 months, dairy kept of nightly wear. Polysomnographic data obtained from one night at the end of three months.
  Interventions: Device: Michigan Bite Splint

INTERVENTIONS:
Device: SOVA Bite Splint — Over-the-counter thermoplastic bite splint blank, heated, molded to fit.
  Arms: SOVA bite splint
Device: Michigan Bite Splint — Heat-cured acrylic bite splint fabricated by dentist/dental technician to fit
  Arms: Michigan Bite Splint

SUMMARY:
Clinical trials of bite splint use and night time tooth grinding have not been performed. Consequently, there are no definitive outcome measures or efficacy standards that can be applied to large clinical trials. The present preliminary trial will determine what objective measures can be used to evaluate efficacy. The outcome variables will fall into four categories: (1) fabrication efficacy, (2) compliance, (3) functional efficacy, and (4) user satisfaction. The immediate goals will: (1) focus on the over-the counter SOVA night guard, (2) conduct tests under controlled clinical conditions using the 'gold standard', the acrylic 'bite splint' or 'orthotic', hereafter called the "Michigan bite splint", to compare the performance and efficacy of the SOVA night guard. Subsequent studies will be able to use the outcome variables identified in this study for broader clinical trials.

Specific Aim 1. To compare the SOVA night guard to the custom-acrylic Michigan bite splint in clinical laboratory conditions. Hypothesis: There will be no significant differences between the devices in terms of fabrication efficacy, functional efficacy or user satisfaction.

Specific Aim 2. To compare the SOVA night guard to the custom-acrylic Michigan bite splint under ecologically relevant conditions, i.e., the home environment. Hypothesis: There will be no significant differences between the devices in terms of compliance or functional efficacy.

DETAILED DESCRIPTION:
Subjects. Sample size estimations are based upon a recent review of randomized clinical trials, in which acrylic appliances were evaluated (see Appendix 2 in (Huynh et al., 2007)). The mean +/- 1 standard deviation (SD) number of bruxism episodes per hour with a Michigan bite splint was 3.97 + 0.58, and for a palatal splint, the mean +/- 1 SD was 4.45 + 0.63. Using these means and the higher SD (0.63), along with an alpha = 0.05 and beta = 0.8, a study would be sufficiently powered with sample sizes of 29 per group. Based on other Michigan studies, wherein recruitment, exclusion and attrition rates are known, it is estimated that an initial screening sample size of 120 will be necessary to end up with 29 per group.

There will be two treatment groups: a group receiving supervised training in the fabrication of the SOVA night guard (SOVA) and a group receiving the Michigan custom-acrylic bite splint (MI BS). Two groups times 29 subjects per group equals 58 total needed for analysis.

Care will be taken to match the randomized groups for age, ethnicity, gender and temporomandibular disorders (TMD) signs/symptoms. Alternatively these will be modeled as nuisance variables if attrition rates create bias or there is a lack of sufficiently sized screening pools.

Screening. Candidates will undergo a screening to assess co-morbidities and to identify inclusion and exclusion criteria. Standard questionnaires and screening instruments and a brief clinical exam will be performed. Subjects meeting the acceptance criteria will be randomly assigned to one of the two groups using stratified randomization procedures (Suresh, 2011). Alginate impressions will be taken, and impressions poured in stone. The models will be used either to fabricate the MI BS or to assess SOVA appliances for fabrication efficacy.

Splint delivery. For the SOVA group, subjects will be asked to fabricate SOVA devices in the clinical laboratory while receiving feedback from trained and calibrated study 'instructors'. Fabrication will use manufacturer instructions. Calibrated instructors will be blinded to the study's objectives, as will subjects. A "Michigan" acrylic bite splint will be fabricated using standard clinical practice and checked for fit and quality on subjects assigned to the MI BS group.

Subjective fabrication assessment. Standardized questionnaires and box scales will be used to assess ease of fabrication, ease of instructions, and other related issues for the devices.

Quantitative fabrication assessments. Four aspects of fabrication will be evaluated by investigators: (1) stability-does the device move independently of the maxilla and is the mandible stabilized by the device, (2) retention-does the device resist displacement, (3) tissue adaptation-how much spacing exists between the maxilla and the device and between the device and mandible, and (4) health of the teeth, gingival, tongue, palate and lips.

Stability and retention will be quantitatively assessed with jaw movement (MaxTraq motion analysis system, Innovision, Columbiaville, MI) and electromyography (EMG) (LabChart, ADInstruments, Colorado Springs, CO) data and force sensors. For position-stability assessment, maxilla, mandible and the splint will be simultaneously recorded from at least three sites to capture 6 degrees of movement freedom. Subjects will clench, grind, perform closed border movements and vacuous chewing (verified with EMG and force sensors). For retention assessment, subjects will perform a series of tests designed to dislodge the device, e.g., tapping, forced blowing, coughing, chewing on gum. Stability and retention indices will be created based on whether device movements vary independently of jaw movements and applied bite forces, and how force sensor output varies during dislodgement exercises. Deviations will be used to form standardized indices of stability and retention, with smaller values representing greater stability and retention. Note that a major part of the study will be to develop the appropriate methods to make these measurements, as it is not clear how this should be done ideally.

Tissue adaptation will be assessed by 3D laser scanner. The occlusal, facial and lingual surfaces of the upper arch will be scanned as will the inner surface of the night guards. An index of adaptation will be developed based on the volumetric spaces separating the teeth from the device, using topological software. Smaller volumes will represent better tissue adaptation. Volumetric indices will be compared between devices via ANOVA or appropriate statistical methods. Note that a major part of this study will be to develop an accurate and precise way of measuring volumetric spacing, as such methods have not yet been developed.

Tissue health will be assessed via appropriate, standard methods currently used in cariology and periodontology clinical studies (Monse et al., 2012; Tirapellia et al., 2010). Baseline measurements will be compared with post-device wear measurements. Between-group differences will be studied with a repeated measures ANOVA or appropriate statistical methods.

Compliance assessment. Compliance assessments will focus on: (1) how often the device is worn, (2) whether the device is removed at inappropriate times during the night, (3) whether alternative devices are used. Compliance will be assessed via subject self-report, nocturnal EMG recording devices and microwear methods. Subjects would be blinded to the purpose of the technological methods. Occlusal microwear patterns are unique to the surfaces against which occlusion occurs, and the microwear changes on a daily basis (Ungar et al., 2003). Hence, microwear assessment should provide definitive evidence of splint compliance. Microwear analysis methods will be developed as part of this study for these purposes.

Functional efficacy. Two questions will be addressed under functional efficacy: (1) does the device alter bruxing activity, and (2) how do the teeth and device hold up under bruxing activity. Some of the technology used for compliance assessment, above, can be used here. Gold standard methods for evaluating bruxing activity rely on polysomnography (PSG) and EMG activity; therefore, it these technologies will be used as well. To address the second question, how do the teeth hold up, 3-D laser scanning technology will be developed and used to measure changes in macroscopic tooth structure, and confocal microscopy and scale-sensitive fractal analysis will be assessed for utility in diagnosing microwear.

User satisfaction. This will be assessed through a series of standardized questionnaires adopted from other clinical studies, e.g., the Oral Health Impact Profile (Slade and Spencer, 1994), the Tampa Scale for Kinesiophobia: TMD (Visscher et al., 2010), the TMD pain screener (Gonzalez et al., 2011). Questionnaires used in the SISU field tests (SISU mouthguards preliminary results), as well as forced choice, box scales and statistical methods developed in another study (Lin, 2008; Lin et al., 2013) will also prove useful for assessment of patient satisfaction. Also questions such as, does the device hurt or pinch anywhere, does your bite feel 'off' when you first remove the guard, etc. will be used to assess specific aspects of user satisfaction.

Repeated measures (Week 1 check-up and 4 Month check-up). Compliance, stability, retention, tissue adaptation and health, functional efficacy and user satisfaction will be assessed two times, viz., 1 week after delivery and 4 months after delivery. This will provide a rigorous data set, reduce subject attrition and thus allow for both publications and further clinical trials to be pursued.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Tooth wear
* Night time grinding and clenching noises
* Full dentition sans 3rd molars
* Ability to follow instructions
* Ability to report to the clinical laboratory at appointed times over the course of the study.

Exclusion Criteria

* Decayed, missing teeth
* Cardiovascular disease
* Sleep apnea, sleep disorders, movement disorders
* Active orthodontics
* Periodontal disease
* Partial or full dentures
* Medications with movement disorders as side effects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-11; Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Gerstner, DDS, MS, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Cunha-Cruz J, Pashova H, Packard JD, Zhou L, Hilton TJ; for Northwest PRECEDENT. Tooth wear: prevalence and associated factors in general practice patients. Community Dent Oral Epidemiol. 2010 Jun;38(3):228-34. doi: 10.1111/j.1600-0528.2010.00537.x. Epub 2010 Mar 29. PMID 20370807
- [Background] Dworkin SF, LeResche L. Research diagnostic criteria for temporomandibular disorders: review, criteria, examinations and specifications, critique. J Craniomandib Disord. 1992 Fall;6(4):301-55. No abstract available. PMID 1298767
- [Background] Fricton J, Look JO, Wright E, Alencar FG Jr, Chen H, Lang M, Ouyang W, Velly AM. Systematic review and meta-analysis of randomized controlled trials evaluating intraoral orthopedic appliances for temporomandibular disorders. J Orofac Pain. 2010 Summer;24(3):237-54. PMID 20664825
- [Background] Gonzalez YM, Schiffman E, Gordon SM, Seago B, Truelove EL, Slade G, Ohrbach R. Development of a brief and effective temporomandibular disorder pain screening questionnaire: reliability and validity. J Am Dent Assoc. 2011 Oct;142(10):1183-91. doi: 10.14219/jada.archive.2011.0088. PMID 21965492
- [Background] Huynh N, Manzini C, Rompre PH, Lavigne GJ. Weighing the potential effectiveness of various treatments for sleep bruxism. J Can Dent Assoc. 2007 Oct;73(8):727-30. PMID 17949541
- [Background] Klasser GD, Greene CS, Lavigne GJ. Oral appliances and the management of sleep bruxism in adults: a century of clinical applications and search for mechanisms. Int J Prosthodont. 2010 Sep-Oct;23(5):453-62. PMID 20859563
- [Background] Lin AI, Braun T, McNamara JA Jr, Gerstner GE. Esthetic evaluation of dynamic smiles with attention to facial muscle activity. Am J Orthod Dentofacial Orthop. 2013 Jun;143(6):819-27. doi: 10.1016/j.ajodo.2013.01.017. PMID 23726332
- [Background] Maeda Y, Kumamoto D, Yagi K, Ikebe K. Effectiveness and fabrication of mouthguards. Dent Traumatol. 2009 Dec;25(6):556-564. doi: 10.1111/j.1600-9657.2009.00822.x. Epub 2009 Sep 24. PMID 19788425
- [Background] Monse B, Duijster D, Sheiham A, Grijalva-Eternod CS, van Palenstein Helderman W, Hobdell MH. The effects of extraction of pulpally involved primary teeth on weight, height and BMI in underweight Filipino children. A cluster randomized clinical trial. BMC Public Health. 2012 Aug 31;12:725. doi: 10.1186/1471-2458-12-725. PMID 22938147
- [Background] Ohrbach R, Larsson P, List T. The jaw functional limitation scale: development, reliability, and validity of 8-item and 20-item versions. J Orofac Pain. 2008 Summer;22(3):219-30. PMID 18780535
- [Derived] Gerstner G, Yao W, Siripurapu K, Aljanabi H, Decker A, Ludkin D, Sinacola R, Frimenko K, Callaghan K, Penoyer S, Tewksbury C. Over-the-counter bite splints: A randomized controlled trial of compliance and efficacy. Clin Exp Dent Res. 2020 Dec;6(6):626-641. doi: 10.1002/cre2.315. Epub 2020 Aug 10. PMID 32779386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 104 individuals screened, 81 met criteria
Pre-assignment Details: 14 individuals dropped out prior to group assignment during consent process due to time/scheduling issues
Groups:
- SOVA Bite Splint: SOVA Bite splint: Over-the-counter, heat-and-mold bite splint. Investigators evaluate subject self-fabrication, and evaluate fit. Subjects wear splint nightly for one week. Polysomnographic data obtained from one night during the week. Subjects continue to wear splint for 4 months, dairy kept of nightly wear. Polysomnographic data obtained from one night at the end of three months.
  SOVA Bite Splint: Over-the-counter thermoplastic bite splint blank, heated, molded to fit.
- Michigan Bite Splint: Michigan bite splint: Gold standard, custom acrylic bite splint made for subjects. Investigators evaluate fit. Subjects wear splint nightly for one week. Polysomnographic data obtained from one night during the week. Subjects continue to wear splint for 4 months, dairy kept of nightly wear. Polysomnographic data obtained from one night at the end of three months.
  Michigan Bite Splint: Heat-cured acrylic bite splint fabricated by dentist/dental technician to fit
Period: Overall Study
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Started | 35 | 32
Clinical Exam, Impressions | 35 | 32
Splint Delivery, Assessments | 33 | 31
1 Week Follow-up, Assessments | 33 | 31
4 Month Follow-up, Assessments | 30 | 31
Completed | 30 | 31
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOVA Bite Splint | Michigan Bite Splint | Total
Number analyzed (Participants) | 35 | 32 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 32 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.5 (3.33) | 25.4 (3.83) | 25.5 (3.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 16 | 17 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 31 | 30 | 61
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 5 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 26 | 23 | 49
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 32 | 67
Bruxing Self-report [Count of Participants; unit: Participants] — 4-point scale reflecting frequency of nights bruxing per week or per month
  Participants
    < 1 night / month | 1 | 0 | 1
    1-3 nights / month | 6 | 4 | 10
    1 -3 nights / week | 15 | 14 | 29
    4 - 7 nights / week | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Nights of Splint Wear for Four Months Per Subject.
Description: Count of the total number of entire nights that subjects wore the splint provided to them in the study.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: nights
Groups:
- SOVA Bite Splint: SOVA Bite splint: Over-the-counter, heat-and-mold bite splint. Investigators evaluate subject self-fabrication, and evaluate fit. Subjects wear splint nightly for one week. Polysomnographic data obtained from one night during the week. Subjects continue to wear splint for 4 months, dairy kept of nightly wear. Polysomnographic data obtained from one night at the end of four months.
  SOVA Bite Splint: Over-the-counter thermoplastic bite splint blank, heated, molded to fit.
- Michigan Bite Splint: Michigan bite splint: Gold standard, custom acrylic bite splint made for subjects. Investigators evaluate fit. Subjects wear splint nightly for one week. Polysomnographic data obtained from one night during the week. Subjects continue to wear splint for 4 months, dairy kept of nightly wear. Polysomnographic data obtained from one night at the end of four months.
  Michigan Bite Splint: Heat-cured acrylic bite splint fabricated by dentist/dental technician to fit
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
nights | 93.6 (31.62) | 98.7 (41.13)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.23, t-test, 2 sided

2. Secondary Outcome: Number of Bruxing Events Per Hour Sleep Per Night.
Description: Polysomnographic monitors were used to evaluate masticatory muscle activity during sleep. Activity of jaw closing muscles found in the cheeks (masseter muscles) occur in bursts, where a burst is taken as evidence for a jaw clench. The total number of bursts recorded during the night was tabulated and then divided by the total hours of sleep. Means presented are based on data gathered on night 122 (4 months of splint wear) and compared with ANOVA.
Time Frame: 4 months
Population: Polysomnographic data were not available from 5 SOVA and 3 Michigan splint subjects due to data corruption. Corruption typically occurs when a subject either removes the device or an electrode while sleeping, or the recorded data are too noisy to analyze due to electronic interference while the subject is asleep.
Measure: Mean (Standard Deviation); unit: muscle bursts / hour
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 25 | 28
muscle bursts / hour | 52.9 (27.15) | 41.5 (25.11)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.045, ANOVA

3. Secondary Outcome: Splint Material Loss / 4 Months.
Description: Splint wear measured in millimeters. The number is negative to reflect the amount lost, e.g., -0.1 = a tenth of a millimeter lost. High-resolution, computer-scanned models of the splint on the delivery date were combined with high-resolution, computer-scanned models of the same splint after 4 months of wear. Sites where teeth contacted the splints were identified, and material loss in these areas was quantified using a computer program designed to quantify differences between two computer models. The measurement represents the difference between the two models, defined by a mean value sampled from a standard-sized area, which was set to be about the size of a tooth cusp (~ 3 millimeters in diameter). Group means were compared with t-tests.
Time Frame: 4 months
Population: Three SOVA subjects and 1 Michigan subject were not included in the analysis, because the scanned models could not be successfully aligned. This was likely due to a warpage of the impressions taken, warpage in the stone models that were scanned, or error in the model scanning process.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 27 | 30
millimeters | -0.20 (0.170) | -0.17 (0.234)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.665, t-test, 2 sided

4. Secondary Outcome: Compliance -- Appliance Removal at Night
Description: Responses to the question, "I frequently remove the splint during the night" with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out at the end of 4 months of splint wear.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Units on a scale | 1.2 (1.40) | 0.8 (1.19)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.249, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Compliance -- Use of Alternative Devices
Description: Responses to the question, "I use an additional splint" with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out at the end of 4 months of splint wear.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Units on a scale | 0.6 (1.30) | 0.5 (1.06)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.626, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Functional Efficacy -- Tooth Wear
Description: Tooth wear measured in millimeters. The number is negative to reflect the amount lost, e.g., -0.1 = a tenth of a millimeter lost. High-resolution, computer-scanned models of the teeth in the lower jaw on the delivery data were combined with high-resolution, computer-scanned models of the same teeth and jaw after 4 months of splint wear. Sites where teeth showed cratering due to dentin exposure were targeted to make these measurements. Changes in these areas was quantified using a computer program designed to quantify differences between two computer models. The measurement represents the difference between the two models, defined by a mean value sampled from a standard-sized area, which was set to be about the size of dentin exposure areas (~ 1 millimeter in diameter). Group means were compared with t-tests.
Time Frame: 4 months
Population: Mandibular models were not available for two SOVA patients.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 28 | 31
millimeters | -.060 (0.013) | -.053 (0.013)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.695, t-test, 2 sided

7. Secondary Outcome: Functional Efficacy -- Alteration of Bruxism Habit, Self Report of Reduced Bruxism
Description: Responses to the question, "The splint helps my bruxism." with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out at the end of 4 months of splint wear.
Time Frame: 4 months
Population: Question not answered by one SOVA participant.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 29 | 31
Units on a scale | 2.7 (1.00) | 3.0 (0.87)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.255, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Functional Efficacy -- Alteration of Bruxism Habit, Self-Report of Muscle Relaxation
Description: Responses to the question, "The splint relaxes my jaw muscles." with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out at the end of 4 months of splint wear.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Units on a scale | 1.9 (0.94) | 2.5 (1.09)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = .049, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: User Satisfaction -- Ease of Fabrication
Description: Responses to the question, "The splint was easy to fabricate" with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out at the end of the appointment during which time the splints were made by participants.
Time Frame: On day of delivery
Population: One SOVA bite splint participant did not respond. Participants with the Michigan bite splint did not fabricate their splints; hence, this question is irrelevant to them.
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 29 | 0
Participants
  Strongly disagree | 1 |
  Somewhat disagree | 3 |
  Neither agree nor disagree | 1 |
  Somewhat agree | 13 |
  Strongly agree | 11 |

10. Secondary Outcome: User Satisfaction -- Ease of Instructions
Description: Responses to the question, "The instructions were easy to follow" with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out at the end of the appointment during which time the splints were made by participants.
Time Frame: On day of delivery
Population: One SOVA bite splint participant did not respond to this question. Michigan bite splint participants did not fabricate their splints; hence, this question was irrelevant for them.
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 29 | 0
Participants
  Strongly disagree | 0 |
  Somewhat disagree | 1 |
  Neither agree nor disagree | 2 |
  Somewhat agree | 16 |
  Strongly agree | 10 |

11. Secondary Outcome: User Satisfaction -- Self-Report of Splint Fit
Description: Responses to the question, "The splint fits well" with a 5-point Likert scale, anchored on the left with "Strongly Disagree" (receiving a score of 0) and on the right with "Strongly Agree" (receiving a score of 4). Question was filled out during the final appointment.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Units on a scale | 3.1 (1.23) | 3.3 (0.83)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.750, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Fabrication Efficacy -- Estimated Bite Forces During Stability Testing
Description: Estimated bite forces in kilograms associated with performing each of the following tasks: moving the jaw in extreme positions with pressure against the splint (Border), clenching (Clench), grinding side to side (Grind Lateral), grinding front to back (Grind Protrusive), tapping hard on splint (Tap). Overall means for each treatment group (SOVA and Michigan splints) are also reported.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
kilograms
  Group Means | 28.4 (1.13) | 16.7 (1.09)
  Border | 24.4 (1.14) | 11.7 (1.11)
  Clench | 49.7 (1.14) | 35.5 (1.11)
  Grind Lateral | 17.7 (1.14) | 10.4 (1.10)
  Grind Protrusive | 25.4 (1.15) | 12.3 (1.11)
  Tap | 34.1 (1.14) | 24.4 (1.11)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p < 0.01, Mixed Models Analysis — The P-value given is the computed value

13. Secondary Outcome: Fabrication Efficacy -- Retention Trials Week 1
Description: Number of times splint was dislodged while performing eight different movements, with each movement being performed five times (maximum number therefore = 40). Dislodgement meant that, after performing the movement, the splint either fell off the teeth completely or that biting down on the splint resulted in its being reseated on the teeth.
Time Frame: 1 week
Population: Data not available for one SOVA participant.
Measure: Mean (Standard Deviation); unit: Occurrences
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 29 | 31
Occurrences | 1.1 (1.93) | 0.6 (1.69)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.544, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Fabrication Efficacy -- Retention Trials, Month 4
Description: as for outcome 13
Time Frame: 4 months
Population: Data not available for one SOVA participant.
Measure: Mean (Standard Deviation); unit: Number of occurrences out of 40.
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 29 | 31
Number of occurrences out of 40. | 1.7 (3.42) | 0.6 (1.86)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.220, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Fabrication Efficacy -- Tissue Adaptation, Palatal Rim. Number of Participants With Poor Adaptation
Description: Palate-side of splints was evaluated for contact with the palate. Splints that were > 1 mm from contact with palate, from molar to molar were graded as 1 (poor adaptation); splints in continuous contact or lacking contact < 1mm with palate, from molar to molar were graded as 0 (good adaptation). Number of participants with splints in each group with poor adaptation is reported.
Time Frame: Day of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Participants | 7 | 2
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.081, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Fabrication Efficacy -- Tissue Adaptation, Facial Rim. Number of Participants With Poor Adaptation
Description: Lip- and cheek-sides of splints were evaluated for contact with the premolar and molar teeth. Splints lacking contact (> 1 mm space between splint and teeth) were graded as 1 (poor adaptation); splints with < 1 mm space between splint and teeth, from molar to molar as 0 (good adaptation). Inter-proximal contacts Number of total participants with splints in each group with poor adaptation is reported.
Time Frame: Day of Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Participants | 4 | 4
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 1.0, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Fabrication Efficacy -- Tissue Adaptation, Number of Subjects Whose Splints Had Excessive Material
Description: Splint rims were evaluated for thickness. Splints requiring modification by the attending dentist to remove excess material were graded as 1 (poor adaptation); splints that did not require removal of excess material were graded as 0 (good adaptation). Number of participants in each group whose splint manifest poor adaptation is reported.
Time Frame: Day of Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Participants | 5 | 4
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.731, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Fabrication Efficacy -- Tissue Adaptation, Tightness. Number of Participants Reporting Excessive Tightness
Description: Splints were evaluated for sensation of tightness on the teeth. SOVA splints that were said to be too tight by the participants and that subsequently required intervention by the attending dentist to fix were graded as 1 (poor adaptation); Michigan splints that were said to be too tight by the participants and that required the attending dentist to spend > 15 minutes of the delivery appointment to fix were graded as 1 (poor adaptation); all splints not meeting these criteria were scored as 0 (good adaptation). Total participants in each group with poorly adapted splints is reported.
Time Frame: Day of Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Participants | 0 | 3
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.238, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Fabrication Efficacy -- Oral Health Plaque Index
Description: The Rustogi et al. Modification of the Navy Plaque Index method of scoring plaque was used. This involves dividing the cheek-facing (Buccal) and the tongue/palate-facing (Lingual) surfaces of each tooth into 9 regions and scoring whether disclosed plaque is present (1) or absent (0) in each of these 9 regions. The total number of regions with plaque was then tabulated as the proportion of total regions for four mouth areas, viz., the cheek sides of the upper teeth (Buccal Upper), the cheek sides of the lower teeth (Buccal Lower), the palate sides of the upper teeth (Lingual Upper) and the tongue sides of the lower teeth (Lingual Lower). Overall means for each treatment group (SOVA and Michigan splints) are also reported.
Time Frame: 1 week and 4 months
Measure: Mean (Standard Deviation); unit: proportion of total regions
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
proportion of total regions
  Buccal Upper, Week 1 | 0.46 (0.187) | 0.42 (0.165)
  Buccal Upper, Month 4 | 0.46 (0.163) | 0.38 (0.155)
  Buccal Lower, Week 1 | 0.41 (0.187) | 0.43 (0.147)
  Buccal Lower, Month 4 | 0.37 (0.135) | 0.39 (0.125)
  Lingual Upper, Week 1 | 0.31 (0.173) | 0.31 (0.174)
  Lingual Upper, Month 4 | 0.29 (0.109) | 0.28 (0.108)
  Lingual Lower, Week 1 | 0.39 (0.127) | 0.44 (0.169)
  Lingual Lower, Month 4 | 0.39 (0.142) | 0.41 (0.138)
  Group Means | 0.39 (0.019) | 0.38 (0.019)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.952, ANOVA — The P-value refers to the difference in group means, see "Group Means" row in the table

20. Secondary Outcome: Fabrication Efficacy -- Oral Health Modified Gingival Index
Description: Gums or gingiva around each tooth is quantified for absence of inflammation (0), mild inflammation around part of the gingiva next to the tooth (1), mild inflammation involving all of the gingiva next to the tooth (2), moderate inflammation (3), or severe inflammation (4). Average scores are created for the cheek side of the upper teeth (Buccal Upper), palate side of upper teeth (Lingual Upper), cheek side of lower teeth (Buccal Lower) and tongue side of lower teeth (Lingual Lower). Mean and standard deviation scores for each of these regions and for week 1 and month 4 are shown as descriptive statistics; statistical results for the between-subject effects are reported. Overall means for each treatment group (SOVA and Michigan splints) are also reported.
Time Frame: 1 week and 4 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 31
Units on a scale
  Buccal Upper, Week 1 | 0.96 (0.628) | 0.92 (0.673)
  Buccal Upper, Month 4 | 1.02 (0.757) | 1.00 (0.747)
  Buccal Lower, Week 1 | 0.87 (0.542) | 0.92 (0.643)
  Buccal Lower, Month 4 | 0.99 (0.713) | 0.95 (0.746)
  Lingual Upper, Week 1 | 0.88 (0.610) | 0.86 (0.67)
  Lingual Upper, Month 4 | 0.95 (0.722) | 0.91 (0.644)
  Lingual Lower, Week 1 | 1.09 (0.679) | 1.03 (0.696)
  Lingual Lower, Month 4 | 1.08 (0.748) | 0.98 (0.726)
  Group Means | 0.93 (0.04) | 0.89 (0.039)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.53, ANOVA — The P-value refers to the difference in group means, see "Group Means" row in the table

21. Secondary Outcome: Stability -- Splint Movement During Jaw Movement Tasks
Description: Movement of each subject's splint on the teeth, due to rocking or dislodgement, measured in millimeters during five repetitions of the following five tasks: clenching, grinding, moving jaw to extreme positions on the splint, tapping, opening maximally. For control, movements of the splint while the jaw was in a rest position (teeth apart, jaw relaxed) were also measured. The maximum movement during the five repetitions of each task was calculated for each subject and used in statistical analyses.
Time Frame: 4 months
Population: Data not available for one participant in the Michigan bite splint treatment group.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 30
millimeters
  Clenching | 0.72 (1.938) | 0.71 (1.583)
  Grinding | 0.83 (1.660) | 0.78 (0.697)
  Border Movements | 0.63 (1.238) | 1.12 (1.331)
  Tapping | 0.33 (0.412) | 0.30 (0.361)
  Maximum Opening | 1.16 (0.940) | 1.60 (1.298)
  Resting | 0.16 (0.177) | 0.22 (0.225)
  Group Means | 0.65 (1.257) | 0.78 (1.143)
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.292, Mixed Models Analysis — The P-value refers to the difference in group means, see "Group Means" row in the table

22. Secondary Outcome: Stability -- Number of Splints Dislodged by Clenching
Description: Count of the number of participants whose individual splints were dislodged at least once when participants clenched their teeth against the splint five times. Numbers are sorted into those that moved < 1 mm, those that moved between 1 - 2 mm, those that moved between 2 - 3 mm and those that moved > 6 mm during the performance of five repeats of clenching. Categories from 3 mm to 6 mm are not included, because no splints fell into this range of values.
Time Frame: 4 months
Population: Data not available for one participant in the Michigan bite splint group
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 30
Participants
  < 1 mm | 26 | 27
  1 - 2 mm | 2 | 1
  2 - 3 mm | 1 | 1
  > 6 mm | 1 | 1
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; The P-value refers to the main effect of treatment group, i.e., differences between SOVA bite splints and Michigan bite splints; Test type: Other; p = 0.289, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Stability -- Number of Splints Dislodged by Grinding
Description: Count of the number of participants whose individual splints were dislodged at least once when participants ground their teeth against the splint to the left (5 times), to the right (5 times, and front to back (5 times). Count is partitioned into those dislodged by < 1 mm, between 1 - 2 mm, between 2 - 3 mm, between 3 - 4 mm, and > 6 mm. Categories between 4 and 6 mm are not included, as no splints fell into this range.
Time Frame: 4 Months
Population: Data not available for one participant in the Michigan bite splint group.
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 30
Participants
  < 1 mm | 26 | 23
  1 - 2 mm | 3 | 4
  2 - 3 mm | 0 | 2
  3 - 4 mm | 0 | 1
  > 6 mm | 1 | 0
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.287, Wilcoxon (Mann-Whitney) — The P-value refers to the main effect of treatment group, i.e., differences between SOVA bite splints and Michigan bite splints

24. Secondary Outcome: Stability -- Number of Splints Dislodged During Border Movement Trials
Description: Count of the number of participants whose individual splints were dislodged at least once when participants performed grinding-like movements of the teeth against the splint in extreme positions. These extreme movements and positions were performed 5 times. Counts are partitioned into those dislodged > 1 mm, those dislodged between 1 - 2 mm, those dislodged 2 - 3 mm, those dislodged 3 - 4 mm, those dislodged 4 - 5 mm, those dislodged 5 - 6 mm and those dislodged > 6 mm.
Time Frame: 4 months
Population: Data not available for one participant in the Michigan bite splint group.
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 30
Participants
  < 1 mm | 28 | 20
  1 - 2 mm | 0 | 5
  2 - 3 mm | 1 | 2
  3 - 4 mm | 0 | 1
  4 - 5 mm | 0 | 1
  5 - 6 mm | 0 | 1
  > 6 mm | 1 | 0
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.505, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 23, analysis 1]

25. Secondary Outcome: Stability -- Number of Splints Dislodged by Tapping
Description: Count of the number of participants whose individual splints were dislodged at least once when participants tapped their teeth on the splint 5 times. Counts are partitioned into the number dislodged < 1 mm, and those dislodged between 1 - 2 mm.
Time Frame: 4 months
Population: Data not available from one participant in the Michigan bite splint group.
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 30
Participants
  < 1 mm | 28 | 28
  1 - 2 mm | 2 | 2
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.643, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 23, analysis 1]

26. Secondary Outcome: Stability -- Number of Splints Dislodged During Maximum Openings
Description: Count of the number of participants whose individual splints were dislodged at least once when participants opened as wide as possible and then closed. The task was repeated five times. Counts are partitioned into the number dislodged < 1 mm, number dislodged between 1 - 2 mm, number dislodged between 2 - 3 mm, number dislodged between 3 - 4 mm and number dislodged between 4 - 5 mm.
Time Frame: 4 Months
Population: Data not available for one participant in the Michigan bite splint group.
Measure: Count of Participants; unit: Participants
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
Number analyzed (Participants) | 30 | 30
Participants
  < 1 mm | 18 | 13
  1 - 2 mm | 7 | 8
  2 - 3 mm | 2 | 2
  3 - 4 mm | 3 | 5
  4 - 5 mm | 0 | 2
Statistical Analysis 1: Comparison: SOVA Bite Splint vs Michigan Bite Splint; Test type: Other; p = 0.923, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 23, analysis 1]

ADVERSE EVENTS:
Time Frame: 4 months
Description: Each participant was followed for four months.
Arm/Group | SOVA Bite Splint | Michigan Bite Splint
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 0/35 | 3/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOVA Bite Splint (N=35) | Michigan Bite Splint (N=32)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Tape sensitivity
Mucosal Bleeding Spot (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Scrape by subject during splint insertion
Tooth Chipped (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT02340663/Prot_SAP_000.pdf